CLINICAL TRIAL: NCT02130050
Title: Metabolic Profiling in Patients With Obstructive Sleep Apnea: From Plasma to Hypoxic Cell Model of Peripheral Monocyte
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201401106RINB
Record Dates: First submitted 2014-04-11; First posted 2014-05-02 (Estimated); Last update posted 2014-05-02 (Estimated); Status verified 2014-04

CONDITIONS: Obstructive Sleep Apnea; Cardiovascular Disease
Keywords: Obstructive Sleep Apnea; Continuous Positive Airway Pressure; Cardiovascular disease; Polysomnography; Metabolomic
MeSH Terms: conditions — Sleep Apnea, Obstructive; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Human plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- OSA Patient: •male patients aged 30 to 65 yr who are newly diagnosed as severe OSA (AHI >=30/hr)
- Control subjects:: •male control subjects are recruited from Heath Check-up Center. Subjects who are matched with OSA patients at age (+/-2 yrs), body height (+/-3cm) and body weight (<100 kg: +/-3kg, >100 kg: +/-4kg) are screened. Only subjects who are not sleepy (ESS<10) and have no OSA (AHI<5/hr PSG)

SUMMARY:
This three-year project aims to

1. Profile the differentially expressed metabolites in healthy patients with severe Obstructive sleep apnea (OSA) before and after six-month continuous positive airway pressure (CPAP) treatment
2. Identify the candidate metabolites involved in biologic pathways attributing to OSA phenotyping and response to CPAP treatment
3. Validate candidate metabolites in the intermittent-hypoxia model of peripheral monocytes

DETAILED DESCRIPTION:
Obstructive sleep apnea is characterized with chronic intermittent hypoxia and sleep fragmentations. The sequels of OSA included excessive daytime sleepiness, cardiovascular disease, and neurocognitive dysfunction which could be reversed with continuous positive airway pressure (CPAP). A couple of biologic pathways have been associated with the phenotyping of OSA which included craniofacial morphology, ventilator control, body fat distribution/metabolism, and sleepiness vulnerability. Metabolomics, a recently developed technique to detect metabolomic profiles, could help to understand the disease pathophysiology and explore biomarkers. So far, only one paper studied the metabolomic profile in patients with OSA where putative identifications of 14 statistically significant features were profiled. Our pilot study comparing the metabolic profiling in OSA patients randomly assigned to therapeutic and subtherapeutic CPAP showed CPAP treatment did alter the metabolomic profile. Seventeen metabolites in three biologic pathways and 13 metabolites in the six biologic pathways were identified in therapeutic and subtherapeutic CPAP, respectively. Sixteen metabolites in three biologic pathways were identified by comparing two groups. However, there were a couple of weakness in studies in the literature and ours. Furthermore, the direct causal relationship of the profiled metabolites and OSA needs to be clarified. Therefore, we plan to compare the metabolic profiling in control subjects and healthy OSA patients, before and after six-month CPAP treatment, to identify candidate metabolites involved in biologic pathways attributing to phenotyping and response to CPAP treatment. Furthermore, candidate metabolites involved in biologic pathways, especially pathways of ROS, inflammation, and metabolism, will be validated in the intermittent hypoxia model of peripheral monocytes.

ELIGIBILITY:
OSA patients

Inclusion Criteria:

* male patients aged 20 to 90 year who have daytime sleepiness (ESS>=10)
* newly diagnosed OSA (AHI>30/hr) by overnight PSG but never been treated

Exclusion Criteria:

* unwilling or unable to perform testing procedure
* past or current smoking history
* medical condition (including cardiovascular disease, chronic pulmonary disease, diabetes, endocrinologic disease, chronic renal failure, and psychiatric disease)
* systemic inflammatory conditions (system lupus erythematosus, rheumatoid arthritis, sarcoidosis, Crohn's disease, and ulcerative colitis)
* active neurologic event
* active infection two weeks prior to screening
* enrolled in other trials in the study period
* other sleep disorders
* sleepy driver
* using maintenance medications

Control subjects

Inclusion Criteria:

* Age-, sex-, body weight-, height-matched subjects with enrolled OSA patients
* non-sleepy
* no OSA confirmed by home sleep study (AHI<5/hr)

Exclusion Criteria:

* unwilling or unable to perform testing procedure
* past or current smoking history
* medical condition (including cardiovascular disease, chronic pulmonary disease, diabetes, endocrinologic disease, chronic renal failure, and psychiatric disease)
* systemic inflammatory conditions (system lupus erythematosus, rheumatoid arthritis, sarcoidosis, Crohn's disease, and ulcerative colitis)
* active neurologic event
* active infection two weeks prior to screening
* enrolled in other trials in the study period
* other sleep disorders
* using maintenance medications

Ages: 20 Years to 90 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: moderate to severe OSA from primary care clinic friends and families from recommendation of OSA patients
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
The expressed metabolites profiles | 6 months
  Profiling the differentially expressed metabolites in control subjects and healthy patients with severe OSA before and after six-month CPAP treatment

SECONDARY OUTCOMES:
Metabolites in the intermittent-hypoxia model of peripheral monocytes | 6 months
  Validate candidate metabolites in the intermittent-hypoxia model of peripheral monocytes

CONTACTS AND LOCATIONS:
Overall Officials: Peilin Lee, M.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan